CLINICAL TRIAL: NCT00907803
Title: Double-Blind, Randomized, Placebo-Controlled, Multi-Center Trial to Assess Safety, Tolerability, and PK of the Anti-Orthopoxvirus Compound ST-246 When Administered as a Single Daily Oral Dose for 14 Days in Volunteers in the Fed State
Brief Title: Safety, Tolerability, Pharmacokinetics (PK) of the Anti-Orthopox Drug, ST-246
Acronym: 246-Safety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SIGA Technologies (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Annie Frimm, Vice President Regulatory Affairs, SIGA Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SIGA-246-004; DMID 08-0055 (Other: NIH Contract: HHSN261002600014C)
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2010-08-27 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Orthopoxviral Disease
Keywords: Orthopoxvirus; Smallpox; This is a safety study only; ST-246 is being studied for treatment of Orthopoxviruses
MeSH Terms: conditions — Smallpox | interventions — tecovirimat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ST-246 400 mg (Experimental): ST-246 400mg (2 x 200 mg Capsules) Orally Once Daily for 14 days
  Interventions: Drug: ST-246 400 mg
- ST-246 600 mg (Experimental): ST-246 600 mg (3 x 200 mg Capsules) Orally Once Daily for 14 days
  Interventions: Drug: ST-246 600 mg
- Placebo (Placebo Comparator): Matching Placebo capsules, Orally Once Daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ST-246 400 mg — Capsules, 400 mg daily for 14 days
  Other Names: Tecovirimat
  Arms: ST-246 400 mg
Drug: ST-246 600 mg — Capsules, 600 mg daily for 14 days
  Other Names: Tecovirimat
  Arms: ST-246 600 mg
Drug: Placebo — Capsules, once daily for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the safety, tolerability, and pharmacokinetics of two clinical doses of the anti-orthopoxvirus drug, ST-246, administered as a single daily oral dose for 14 days to healthy, fed volunteers. The results of this trial determine which dose will be used in expanded pivotal safety trials.

DETAILED DESCRIPTION:
This study is a Phase II, double-blind, randomized, placebo-controlled, multi-center (3 sites) trial to assess the safety, tolerability, and pharmacokinetics of 400 mg and 600 mg Form I ST-246 when administered as a single daily oral dose for 14 days to 107 healthy, fed volunteers between 18 and 74 years of age. Safety parameters included adverse events, vital signs, physical examinations, laboratory tests (hematology, blood chemistry, and urinalysis) and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 75 yrs
2. Healthy volunteer
3. Ability to consent
4. Available for clinical follow-up for study
5. Not taking other medications
6. Adequate venous access
7. Using adequate birth control; negative pregnancy test
8. Able and willing to avoid alcohol for screening and study duration

Exclusion Criteria:

1. Inability to swallow study medication
2. Pregnant or breast-feeding
3. Medical condition, e.g., asthma, hypertension, angioedema, traumatic brain injury other than concussion, bleeding disorder, blood dyscrasia, idiopathic seizures, cardiac disease that limits activity, diabetes, active malignancy, Hepatitis B or C, HIV or AIDS, chronic microbial infection,
4. History of drug allergy that contraindicates study participation
5. Medical, psychiatric, social, occupational or other reason that jeopardizes the safety/rights of participant or renders he/she unable to comply with the protocol (including drug or alcohol abuse, or homelessness)
6. Clinically abnormal ECG
7. Has or will participate in a clinical trial or experimental treatment within 30 days of, or during, the study
8. Cannot or will not do physical exercise 24 hrs before and after PK days
9. Will not consume grapefruit/grapefruit juice during study
10. Vaccination within 2 wks of screening, or planned before Day 42 of study
11. Treatment with prednisone or equivalent immunosuppressant/modulatory drug <3 mths before screening
12. Clinically significant physical exam and lab results <2weeks from 1st study drug dose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center; Erik Ross, MD, Principal Investigator — Apex Research Institute; Jon Ruckle, MD, Principal Investigator — Hawaii Clinical Research Center
Locations (3):
- United States (3):
  - Apex Research Institute, Santa Ana, California
  - Orlando Clinical Research Center, Orlando, Florida
  - Hawaii Clinical Research Center, Honolulu, Hawaii

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at three sites: Apex Research Institute, Santa Ana, CA, Hawaii Clinical Research Center, Honolulu, HI, and Orlando Clinical Research Center, Orlando, FL. The study was conducted in male and female volunteers ages 18 - 75 years inclusive from the sites' databases.
Pre-assignment Details: Following an up to 14-day Screening Period, eligible subjects were randomly assigned to receive either ST-246 400 mg (n=45) or ST-246 600 mg (n=46) or placebo (n=16). Treatment was orally administered after a light meal over a 14-day Treatment Period. There was a 28-day Follow-up Period.
Groups:
- ST-246 400 mg: 400 mg ST-246 (2 x 200 mg capsules) given as a single daily oral dose to 45 subjects for 14 days.
- ST-246 600 mg: 600 mg ST-246 (3 x 200 mg capsules) given as a single daily oral dose to 46 subjects for 14 days.
- Placebo: Matching Placebo capsules given as a single daily oral dose to 16 subjects for 14 days.
Period: Overall Study
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Started | 45 | 46 | 16
Completed | 42 | 43 | 16
Not Completed | 3 | 3 | 0
Not completed — Withdrawal of consent - long commute | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo | Total
Number analyzed (Participants) | 45 | 46 | 16 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 0 | 2
  Between 18 and 65 years | 41 | 40 | 13 | 94
  >=65 years | 2 | 6 | 3 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 41.3 (15.22) | 43.7 (15.81) | 42.5 (17.03) | 42.5 (15.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 9 | 58
  Male | 18 | 24 | 7 | 49
Region of Enrollment [Number; unit: participants]
  United States | 45 | 46 | 16 | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants Who Tolerated a Single Daily Oral ST-246 Dose as Determined by Safety Parameter Changes According to the DAIDS (Division of Acquired Immunodeficiency Syndrome) Adverse Events (AE) Grading Table.
Description: Subjects were administered a single, daily oral dose of ST-246 (400 or 600 mg)and changes in safety parameteres were monitored. Safety parameters included adverse events, vital signs, physical examinations, laboratory tests (hematology, blood chemistry, and urinalysis) and electrocardiograms. The DAIDS AE grading table is a list of common terms and severity (intensity) of parameters used to describe adverse events occurring in NIAID-sponsored clinical studies/trials.
Time Frame: Days 1 to 14; then 24, 48, 72, 96 and 120 hours and 4 weeks after final dose
Population: As per protocol. During the study, a total of 6 withdrawals occurred. These were due to adverse events (2) and consent withdrawal (1) in the 400 mg group, and subject request (1), lost to follow-up (1) and protocol violation (1) in the 600 mg group.
Measure: Number; unit: Participants
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 16
Participants | 34 | 38 | 15

2. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Cmax
Description: Cmax: Maximum drug concentration in plasma determined directly from individual concentration-time data
Time Frame: Day 1 post-dose
Population: As per protocol. All 16 subjects in the placebo group were excluded from the PK population. In addition, 2 subjects in each of the ST-246 400 mg and 600 mg groups were excluded due to early withdrawals.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Number analyzed (Participants) | 43 | 44 | 0
ng/mL | 1170 (429) | 1467 (626) |

3. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Cmax
Description: Cmax: Maximum drug concentration in plasma determined directly from individual concentration-time data
Time Frame: Day 14 post-dose
Population: As per protocol. All 16 subjects in the placebo group were excluded from the PK population. In addition, 4 subjects in each of the ST-246 400 mg and 600 mg groups were excluded from PK analysis due to withdrawals or because PK data fell below the limit of quantitation (BLQ).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Number analyzed (Participants) | 41 | 42 | 0
ng/mL | 1286 (449) | 1523 (607) |

4. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Tmax
Description: Tmax: Time to reach maximum drug concentration in plasma calculated from [plasma] versus time profiles
Time Frame: Day 1 post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Number analyzed (Participants) | 43 | 44 | 0
hours | 4 (1) | 4 (1) |

5. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Tmax
Description: Tmax: Time to reach maximum drug concentration in plasma calculated from [plasma] versus time profiles
Time Frame: Day 14 post-dose
Population: As per protocol. All 16 subjects in the placebo group were excluded from the PK population. In addition, 4 and 5 subjects in the ST-246 400 mg and 600 mg groups respectively, were excluded from PK analysis due to withdrawals or because PK data fell below the limit of quantitation (BLQ).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Number analyzed (Participants) | 41 | 41 | 0
hours | 4 (1) | 3 (1) |

6. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: AUCtau
Description: AUCtau: Area under the plasma concentration-time curve for each dosing interval (from time 0 to 24 hours sample) determined using the linear trapezoidal rule
Time Frame: Day 1 post-dose
Population: As per protocol. All 16 subjects in the placebo group were excluded from the PK population. In addition, 23 subjects in each of the ST-246 400 mg and 600 mg groups were excluded from PK analysis due to early withdrawals or because PK data fell below the limit of quantitation (BLQ) before the 24-hour dosing interval was complete.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 0
ng*hr/mL | 11329 (4945) | 13895 (5702) |

7. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: AUCtau
Description: as for outcome 6
Time Frame: Day 14 post-dose
Population: As per protocol. All 16 subjects in the placebo group were excluded from the PK population. In addition, 5 and 6 subjects in the ST-246 400 mg and 600 mg groups respectively, were excluded from PK analysis due to withdrawals or because PK data fell below the limit of quantitation (BLQ).
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Number analyzed (Participants) | 40 | 40 | 0
ng*hr/mL | 12026 (4255) | 14791 (5712) |

8. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: t½
Description: t½: Observed terminal elimination half-life determined after the last dose on Day 14
Time Frame: Day 14 post-dose
Population: As per protocol. All 16 subjects in the placebo group were excluded from the PK population. In addition, 21 and 20 subjects in the ST-246 400 mg and 600 mg groups respectively, were excluded from PK analysis due to early withdrawals or because PK data fell below the limit of quantitation (BLQ).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Number analyzed (Participants) | 24 | 26 | 0
hours | 26 (11) | 24 (15) |

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Study drug was administered once a day to each dosing group for 14 days, and subjects were followed for an additional 28 days. AEs were recorded throughout this time period.
Arm/Group | ST-246 400 mg | ST-246 600 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/46 | 0/16
Other Adverse Events (participants affected / at risk) | 11/45 | 8/46 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST-246 400 mg (N=45) | ST-246 600 mg (N=46) | Placebo (N=16)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 5 (5) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must obtain the sponsor's written consent to publish any study results and must notify the sponsor within 30 working days prior to publishing.